CLINICAL TRIAL: NCT00431301
Title: Genetic and Environmental Risk Factors for PSP
Brief Title: Risk Factors for Progressive Supranuclear Palsy (PSP)
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1R01AG024040-01A2 (NIH); 1R01AG024040-01A2 (NIH)
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Progressive Supranuclear Palsy
Keywords: Progressive Supranuclear Palsy; Epidemiology; Case-Control; Genetic; Environmental; Neurodegenerative Disease; Movement Disorders; Atypical Parkinsonism; Parkinson Plus; Steele-Richardson-Olszewski; PSP
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA will be used for genotyping specific genes of interest related to the disease.

GROUPS / COHORTS (2):
- Case: PSP Cases
- Control: Healthy Controls

SUMMARY:
Progressive supranuclear palsy (PSP) is the most common atypical parkinsonian movement disorder. This study will determine the role of specific genetic, occupational and environmental components in the development of PSP by evaluating patients with this disorder and age and gender matched controls.

DETAILED DESCRIPTION:
This proposal will determine: (1) if there is an association between PSP and specific genes of interest; (2) if there is an association between PSP and occupational and/or environmental chemical exposures functionally or structurally similar to known parkinsonian toxicants; and (3) if hypertension or traumatic brain injury prior to symptom-onset is associated with PSP. To disentangle the complex etiology of PSP, this case-control multicenter study involves 500 PSP cases, 500 age/gender matched primary controls, and 500 secondary controls for genetic confirmation. Understanding the etiology of PSP may also help explain the causes of other related diseases such as Alzheimer's disease. This multidisciplinary team of movement disorder specialists, epidemiologists, geneticists, biostatisticians, industrial hygienist and toxicologist is well suited to unravel the etiology of PSP.

ELIGIBILITY:
Inclusion Criteria:

* PSP patients able to visit one of the screening sites for diagnostic confirmation and able to participate in a one hour telephone interview

Exclusion Criteria:

* No other major neurological disorders
* Unable to communicate by telephone

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with clinically diagnosed Progressive Supranuclear Palsy and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 942 (Actual)
Dates: Start 2006-08; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Litvan, M.D., Principal Investigator — University of Louisville
Locations (10):
- United States (9):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - UCLA, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Emory College of Medicine, Atlanta, Georgia
  - Rush University, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Case Western University, Cleveland, Ohio
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Kelley KD, Checkoway H, Hall DA, Reich SG, Cunningham C, Litvan I. Traumatic Brain Injury and Firearm Use and Risk of Progressive Supranuclear Palsy Among Veterans. Front Neurol. 2018 Jun 20;9:474. doi: 10.3389/fneur.2018.00474. eCollection 2018. PMID 29973911
- See also: PSP study information website — http://www.PSPstudy.com